CLINICAL TRIAL: NCT01696292
Title: Evaluation of Mental Flexibility Through Language Tests in Adolescents With Frontal Brain Damage and in Healthy Children in Ages 8-17
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-04-3435-JL-CTIL
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Persons With Frontal Lobe Damage With no Specific Language Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to shed light on the theoretical concept of mental flexibility and its manifestation in adolescents following frontal lobe damage, and to develop a test battery for young Hebrew speakers.

ELIGIBILITY:
Inclusion Criteria:

* frontal lobe damage
* at least one year after injury
* native hebrew speaker

Exclusion Criteria:

* specific language disorder
* premorbid learning disability

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A group of children ages 8-17 with frontal lobe damage, who are treated at the children rehabilitation center at sheba medical center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children Rehabilitation Department Sheba Medical Center, Ramat Gan, Israel